CLINICAL TRIAL: NCT04309539
Title: - Efficacy of Combined Lateral Femoral Cutaneous Nerve Block With Pericapsular Nerve Group Block Versus Fascia Iliaca Block in Proximal Femoral Fractures
Brief Title: Which Analgesia is Better for Proximal Femoral Fractures?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MFM-IRB, MD.20.02.280
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Proximal Femur Fracture
MeSH Terms: conditions — Proximal Femoral Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia iliaca block (Active Comparator): Patients will receive Fascia iliaca block
  Interventions: Procedure: Fascia iliaca block
- combined LFCN block with PENG block (Active Comparator): Patients will receive a combined lateral femoral cutaneous nerve block with pericapsular nerve group block
  Interventions: Procedure: combined LFCN block with PENG block

INTERVENTIONS:
Procedure: Fascia iliaca block — A linear probe will be placed in the sagittal plane to the inguinal ligament to obtain an image of "bow-tie sign" formed by the muscle fascias, a spinal needle will be inserted 1 cm cephalad Using an in-plane approach, the fascia iliaca is penetrated, 30 mL of bupivacaine 0.25% before spinal anesthesia.
  Arms: Fascia iliaca block
Procedure: combined LFCN block with PENG block — With the patient supine, the linear probe is placed parallel to the inguinal ligament. LFCN appear as a hypoechoic oval structure between the tensor fascia lata and Sartorius muscles. The needle is inserted in plane. 5 mL of LA is injected. The PENG block will be performed in the supine position. A curvilinear probe will be placed transversely over the anterior inferior iliac spine and then rotated counterclockwise 45 degrees. the ilio pubic eminence, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle will be observed. A spinal needle will be inserted in plane to the plane between the psoas tendon and the pubic ramus. 25 mL of bupivacaine 0.25% will be injected
  Arms: combined LFCN block with PENG block

SUMMARY:
This patient population is typically elderly and frail. They are at risk of adverse effects secondary to inadequate pain management such as prolonged admissions and poor functional outcomes.

Regional analgesia is preferred due to their opioid-sparing effects and reduction in related adverse effects but The analgesia from these blocks is only moderate and literature suggests that the obturator nerve (ON) is not covered.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of combined lateral femoral cutaneous nerve block with pericapsular nerve group block versus fascia iliaca block for proximal femur surgery.

Fascia iliaca compartment block is a simple technique to manage pain before positioning for spinal anesthesia performance and it constitutes a practical choice for perioperative pain control.

A recent anatomical study confirmed the innervation of the anterior hip by these 3 main nerves, but also found that the AON and FN play a greater role in the anterior hip innervation than previously reported The high articular branches from FN and AON are consistently found between the anterior inferior iliac spine (AIIS) and the iliopubic eminence (IPE), whereas the ON is located close to the inferomedial acetabulum.

The ultrasound-guided technique for blockade of these articular branches to the hip, the PENG (Pericapsular Nerve Group) block reported significantly reduced pain scores compared with baseline. Roy et al 2019 recommended the use of PENG block together with LFCN block as adjunctive to cover the lateral surgical incision.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I, II and III.

Exclusion Criteria:

* Patient refusal.
* Neuromuscular diseases
* Hematological diseases
* Bleeding abnormality
* Coagulation abnormality.
* Psychiatric diseases.
* Local skin infection at the site of the block.
* Local skin sepsis at the site of the block
* Known intolerance to the study drugs.
* Body Mass Index > 40 Kg/m2.
* Multiple trauma patients.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Time of performance of Spinal Anesthesia | just before surgery.
  Is defined as the time measured from the start of positioning to the completion of the intrathecal bupivacaine injection

SECONDARY OUTCOMES:
Pain measurement at rest | immediately and 1 hour at PACU, then in the surgical ward at 2,4,6,8,12,18 and 24 h after surgery.
  10-cm visual analog scale (VAS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain
Pain measurement on movement | immediately and 1 hour at PACU, then in the surgical ward at 2,4,6,8,12,18 and 24 h after surgery.
  (attempted hip flexion to 15 degrees).: 10-cm visual analog scale (VAS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain
Pain measurement during positioning for spinal anesthesia | Just before surgery
  visual analog scale (0-10, 0: no pain, 10: worst pain imaginable) during changing position from supine to sitting one
The severity of postoperative pain at rest | immediately and 1 hour at PACU, then in the surgical ward at 2,4,6,8,12,18 and 24 h after surgery.
  10-cm visual analog scale (VAS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain
The severity of postoperative pain on movement | immediately and 1 hour at PACU, then in the surgical ward at 2,4,6,8,12,18 and 24 h after surgery.
  (attempted hip flexion to 15 degrees): 10-cm visual analog scale (VAS) for pain, where 0 is equal to no pain and 10 indicates the worst possible pain
Time to onset of Sensory blockade | evaluated 15 and 30 min after block administration
  cold perception loss in the lateral, anterior and medial part of the thigh (corresponding to lateral femoral cutaneous (LFC), femoral (F) and obturator (O)nerve sensory distributions, respectively)
Time to onset of motor block | evaluated 15 and 30 min after block administration
  defined as assessment of quadriceps femoris muscle strength by straight leg raise test to 15 degree and classified as follow: +ve =normal power, -ve =motor weakness
Duration of sensory block | postoperative 24 hours
  blockade is defined as the interval between end of injection and complete end of sensory block (score=2)
Duration of motor block | postoperative 24 hours
  blockade is defined as the interval between end of injection and complete end of injection and complete recovery of normal motor function (score=0),
Anesthesiology satisfaction for patient positioning | just before surgery
  evaluated as 0=unsatisfactory, 1=satisfactory, 2=good or 3=optimal
heart rate | pre-block, 15, 30 min after block, immediately after spinal anesthesia, 5min, 15min then every 30 min till end of surgery
  Changes in heart rate
Mean arterial blood pressure | pre-block, 15, 30 min after block, immediately after spinal anesthesia, 5min, 15min then every 30 min till end of surgery
  Changes in Mean arterial blood pressure
Peripheral oxygen saturation | pre-block, 15, 30 min after block, immediately after spinal anesthesia, 5min, 15min then every 30 min till end of surgery
  Changes in peripheral oxygen saturation as measured with pulse oximetry
Time for first analgesic request | Within 24 hours after surgery
  defined as the time period from end of injection to the first time patient requests analgesia postoperatively
Total analgesics received | for 24 hrs after surgery
  cumulative consumption of opioids during the first postoperative day
Pruritis | Within 24 hours after surgery
  number of patients with pruritis
nausea | Within 24 hours after surgery
  number of patients with nausea
vomiting | Within 24 hours after surgery
  number of patients with vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Mona A Hasheesh, MD, Study Chair — Professor of Anesthesia and Surgical Intensive care,,P; Eiad A Ramzy, MD, Study Director — Associate Professor of Anesthesia and Surgical Intensive care,
Locations (1):
- Mansoura University, emergency hospital, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Yes, Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after completing the study and being accepted for publication.
Access Criteria: The data will be accessible to the investigators and PRS administrators with hiding the identifiers for the patients